CLINICAL TRIAL: NCT03225859
Title: Pilot Test of a Self-Management Program for Completers of Trauma-Focused Therapy
Brief Title: A Self-Management Program for Completers of Trauma-Focused Therapy for PTSD
Acronym: EMPOwER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Syracuse VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2525-P; 1I21RX002525-01A1 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stress Disorders, Posttraumatic; Self-Management
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: The study non-randomized, open-trial pilot test of the intervention with twelve Veterans who will all receive the study intervention.
Masking Description: As everyone in the study will receive the same intervention, no masking is being employed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-Management Program (Experimental): Patients in this arm will receive the therapist assisted self-management intervention following completion of trauma-focused therapy for PTSD.
  Interventions: Behavioral: Self-Management Program

INTERVENTIONS:
Behavioral: Self-Management Program — This therapist-assisted self-management program will increase Veterans' self-efficacy for managing their PTSD, enable the maintenance or building upon gains made in trauma-focused therapy, and encourage engagement in meaningful activities. Patients will have four contacts with their providers over the ten weeks following trauma-focused therapy completion. The intervention will help patients: 1)self-monitor symptoms, 2) continue to practice skills learned in trauma-focused therapy, 3) acquire and apply additional coping skills, 4) engage in meaningful activities, and 5) set goals

SUMMARY:
Veterans who complete trauma-focused therapies (TFTs) report improvements in posttraumatic stress disorder symptoms, quality of life, and social and role functioning. However, many also report uncertainty regarding their ability to maintain and build upon progress made during TFTs following the end of treatment. Veterans who recently completed a course of TFT believe the likelihood of their ongoing success would be bolstered by mental health services that support additional practice and reinforcement of skills learned in TFT. Currently no evidence-based approach for post-TFT care exists; however, Veterans' reported treatment needs are well-suited to a therapist-assisted self-management approach. The objective of this project is to complete Stage 1 (intervention refinement and piloting) of the Stage Model of Treatment Development for a post-TFT therapist-assisted self-management program designed to help Veterans maintain or build upon gains made in TFT, increase self-efficacy for managing their PTSD symptoms, and enhance community engagement. The aims of the project are to: 1) Refine a self-management treatment protocol through eliciting feedback from experienced TFT providers on a draft of the self-management program, 2) Conduct a pilot open trial to assess the acceptability and feasibility of the self-management program, and 3) Explore the effects of the program on Veterans' confidence in managing their PTSD and Veterans' functioning, quality of life, community engagement, and mental health symptoms.

DETAILED DESCRIPTION:
Impact: Findings from this project will improve the mental health and well-being of Veterans with posttraumatic stress disorder (PTSD) by refining and evaluating the first post-trauma focused therapy (TFT) intervention designed to help Veterans increase self-efficacy for managing their PTSD symptoms, maintain or build upon gains made in TFT, and increase community engagement. The current VA / Department of Defense PTSD clinical practice guidelines recommend decreasing the frequency and intensity of care (e.g. stepping-down) following successful TFT completion; this project is the initial step in developing the first evidence-based intervention for this important process. The project will advance RR&D's missions of evaluating interventions designed to maximize psychological recovery and prioritizing functional outcomes and societal engagement. Finally, the project will advance the scientific literature by being the first examination of a self-management intervention designed to be used to step down from an intensive course of therapy for PTSD.

Background: TFTs reduce the suffering associated with PTSD; a majority of Veterans who complete prolonged exposure or cognitive processing therapy report improvements in PTSD symptomology, quality of life, and functioning. Despite their effectiveness, emerging data suggest that Veterans who complete TFTs continue to perceive a need for mental health treatment; the investigators' pilot data demonstrated that the primary post-TFT mental health treatment need among completers who experienced at least a partial improvement in PTSD symptoms is support for additional practice and reinforcement of skills learned in TFT. Veterans expressed low self-efficacy for maintaining or building upon their existing gains and believed continued contact with their TFT therapist would increase their likelihood of success. These treatment needs are particularly well-suited to a therapist-assisted self-management approach. Self-management protocols teach patients to be responsible for the day-to-day management of their symptoms, thereby emphasizing patients' roles in wellness. The existing literature on self-management interventions for PTSD has demonstrated that such approaches are acceptable, safe, and effective; however, they have exclusively been used as stand-alone treatments or as the first step up in a stepped-care model. Therefore, the investigators are proposing the first examination of a self-management intervention designed to be used to step down from an intensive course of TFT for PTSD.

Objectives: The objective of this study is to complete stages 1A and 1B of the Stage Model of Treatment Development for the self-management program for Veterans who have recently completed a course of TFT for PTSD. Specifically, the investigators will: (1) Refine a self-management treatment protocol through eliciting feedback from experienced TFT providers, (2) Conduct a pilot open trial to assess the (a) acceptability of the self-management program components, structure, and materials and (b) feasibility of the self-management program (retention and intervention fidelity) and study approach (screening, recruitment, assessment process), and (3) Explore the effects of the program on Veterans' confidence in managing their PTSD (self-efficacy), functioning, quality of life, community engagement, and mental health symptoms.

Methods: To achieve Aim 1, the investigators will conduct semi-structured individual interviews with a sample of TFT providers (n = 10-12), during which participants will be asked to provide feedback on the planned components and structure of the self-management program. To achieve Aims 2 and 3, the investigators will enroll twelve Veterans in a non-randomized, open-trial pilot test of the intervention at the Minneapolis VA Healthcare Systems (VAHCS). Enrolled Veterans will complete survey batteries immediately post-TFT, and survey batteries and qualitative interviews two weeks after the final self-management program therapist contact. Findings from this project will strongly position us to apply for Merit funding to conduct a randomized clinical trial (Stage 2 of the Stage Model of Treatment Development) of this innovative self-management program.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate if they:

* completed a course of individually-delivered trauma-focused therapy (TFT) with a provider trained to deliver the self-management intervention at the Minneapolis VAMC
* experienced a clinically meaningful reduction in PTSD symptomology (PCL decrease of at least 10 points) from pre-TFT to the time of the enrollment
* at the time of enrollment are not planning to initiate another active course of psychotherapy for PTSD in the following three months
* are willing to participate in a self-management intervention, and
* can provide informed consent

Exclusion Criteria:

* Veterans will be excluded if they have suicidal or homicidal ideation that in the opinion of their TFT therapist needs to be the focus of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M. Kehle-Forbes, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Research datasets included in primary publications resulting from this proposed research will involve large amounts of individual PHI data and cannot reasonably or efficiently be fully deidentified. Investigators will create analytic datasets that can be requested by outside investigators. These data however will remain within the VA firewall and be housed on VINCI data servers. Outside investigators can follow VA procedures and receive training and approval for access within VA firewalls.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We identified 23 eligible patients. Twelve (52%) veterans enrolled, five (22%) declined participation, five (22%) were eligible but not contacted because they were not identified prior to their final PE/CPT session, and one (4%) veteran was unreachable. Eighty Veterans who were not eligible for EMPOWER were also identified in our screening procedures; failure to complete PE/CPT (n = 41; 51%) and participation in co-occurring studies (n = 12; 29%) were the most common reasons for exclusion.
Period: Overall Study
Arm/Group | Self-Management Program
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Self-Management Program
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants] — Population: Participant age not collected for this study.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Service Era [Count of Participants; unit: Participants] — Categorical Military Service Era
  Participants
    Iraq & Afghanistan Veterans | 9
    Gulf War 1/Post-Vietnam Era Veterans | 1
    Vietnam Veterans | 2

OUTCOME MEASURES:

1. Primary Outcome: Credibility-Expectancy Scale (Credibility Subscale)
Description: Measures treatment rationale credibility in clinical outcome studies (range 1-9; higher scores = higher credibility).
Time Frame: Prior to first self-management session (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 12
score on a scale | 6.39 (1.73)

2. Primary Outcome: Client Satisfaction Scale
Description: Measures client satisfaction with mental health services (range = 8-32; higher scores = higher satisfaction)
Time Frame: Three months after first self-management session (follow-up)
Population: Includes the 9 patients who provided data for this post-treatment assessment timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 9
score on a scale | 29.67 (2.74)

3. Secondary Outcome: Change From Baseline in Illness Perception Questionnaire - Revised (Personal Control Subscale)
Description: Measures patients' self-efficacy for managing PTSD symptoms; range = 1-5 (higher scores = greater perceived control; change from pre- to post-intervention reported.
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Data from all participants who completed the post-treatment survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 9
score on a scale | 0.33 (1.66)

4. Secondary Outcome: Change From Baseline on PTSD Checklist - 5
Description: Measures DSM-5 PTSD symptoms; Range = 0-80; higher scores = more severe symptoms; change score from pre- to post-treatment reported
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Data reported for all participants who completed post-treatment survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 9
score on a scale | -1.67 (8.26)

5. Secondary Outcome: Change From Baseline on Patient Health Questionnaire - 9
Description: Measures symptoms of depression; range = 0-27; higher scores = more severe symptoms; pre- to post-treatment change score reported
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Participants who provided complete data in post-treatment survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 7
score on a scale | -0.14 (2.79)

6. Secondary Outcome: Change From Baseline on Recovery Orientation Scale (Current Mental Health Subscale)
Description: Measures patients' perceived mental health; range 1-5; lower scores = better perceived mental health
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Data reported for all participants who provided complete post-treatment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 7
score on a scale | -1.0 (0.64)

7. Secondary Outcome: Change From Baseline on World Health Organization Quality of Life - BREF
Description: Measures patients' current quality of life; higher score = better quality of life; range = 0-100. Change score from pre- to post-treatment reported
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Data for all participants who provided complete post-treatment survey data
Measure: Mean (Standard Deviation); unit: Change of score on scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 8
Change of score on scale | 6.62 (6.25)

8. Secondary Outcome: Change From Baseline on Military to Civilian Questionnaire
Description: Measures patients' community engagement; range: 0-4; higher scores = more difficulty; change score from pre- to post-intervention reported
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Data from participants who provided complete post-treatment survey data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 9
score on a scale | -0.27 (0.41)

9. Secondary Outcome: Change From Baseline on Brief Inventory of Psychosocial Functioning
Description: Measure of PTSD-related psychosocial functional impairment; higher scores = more severe; range = 0-49; change from pre- to post-treatment reported
Time Frame: Prior to first self-management session (baseline) and three months after first self-management session (follow-up)
Population: Data for participants who provided complete post-treatment survey data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-Management Program
Number analyzed (Participants) | 9
units on a scale | 4.44 (14.02)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Self-Management Program
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Self-Management Program (N=12)
Hospitalization (Cardiac disorders) | 1 — Participant presented to the ER with cardiac concerns and was hospitalized. This was unanticipated and can not be determined to be directly related to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03225859/Prot_SAP_000.pdf